CLINICAL TRIAL: NCT02061514
Title: The Effect of Two Different General Anesthesia Regimes on Postoperative Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor in Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SLEEP_ANNIE
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia; Surgery; Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Maintenance; Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- maintenance with desflurane (Experimental): in patients allocated to the desflurane group, general anesthesia will be maintained with desflurane
  Interventions: Procedure: maintenance with desflurane
- maintenance with propofol (Active Comparator): in patients allocated to the propofol group, general anesthesia will be maintained with propofol
  Interventions: Procedure: maintenance with propofol

INTERVENTIONS:
Procedure: maintenance with desflurane — in patients allocated to the desflurane group, general anesthesia will be maintained with desflurane
  Arms: maintenance with desflurane
Procedure: maintenance with propofol — in patients allocated to the propofol group, general anesthesia will be maintained with propofol
  Arms: maintenance with propofol

SUMMARY:
* Major surgery can lead to postoperative disturbances in sleep patterns with subjective deterioration of sleep quality according to patients' reports as well as objective alterations of sleep architecture, as recorded by polysomnography
* Factors implicated in postoperative sleep disturbances include but are not limited to the severity of the surgical procedure, the neuroendocrine response to surgery, inadequate treatment of postoperative pain and external factors interfering with sleep, such as light, noise and therapeutic procedures
* There are differences in the molecular mechanisms inhalational anesthetics and intravenous agents affect different brain regions to induce anesthesia. Our hypothesis is that these differences may also be evident during the postoperative period, affecting brain functions which are involved in postoperative sleep architecture. So, the aim of this study will be to assess the effect of two different anesthetic techniques (propofol versus desflurane) of maintaining general anesthesia in patients subjected to similar major operations
* Patients will be assessed with the Pittsburgh Sleep Quality Questionnaire (PSQI), regarding preoperative and long term postoperative sleep quality, sleep diaries regarding early postoperative sleep quality and biochemical markers (cortisol, prolactin and melatonin) regarding neuroendocrine response to surgery and disturbances in endogenous circadian secretion associated with sleep

DETAILED DESCRIPTION:
* Major surgery can lead to postoperative disturbances in sleep patterns with subjective deterioration of sleep quality according to patients' reports as well as objective alterations of sleep architecture, as recorded by polysomnography
* These disturbances include severe sleep fragmentation, rapid eye movement (REM) and slow wave sleep significant reductions in duration as well as an increase in non-REM sleep stages. Spontaneous awakenings are also frequently reported
* After the third or fourth postoperative day, there is a substantial rebound in total REM activity, with frequent reports of vivid nightmares
* Factors implicated in postoperative sleep disturbances include but are not limited to the severity of the surgical procedure, the neuroendocrine response to surgery, inadequate treatment of postoperative pain and external factors interfering with sleep, such as light, noise and therapeutic procedures
* There are differences in the molecular mechanisms inhalational anesthetics and intravenous agents affect different brain regions to induce anesthesia. Our hypothesis is that these differences may also be evident during the postoperative period, affecting brain functions which are involved in sleep architecture, since sleep is an altered state of consciousness like anesthesia. So, the aim of this study will be to assess the effect of two different anesthetic techniques of maintaining general anesthesia in patients subjected to similar major operations
* Patients taking part in the study will be evaluated regarding their preoperative sleep quality by the Pittsburgh Sleep Quality Questionnaire (PSQI). The PSQI examines seven components of sleep quality retrospectively over a period of four weeks: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. The patient self-rates each of these seven areas of sleep. Scoring of answers is based on a 0-3 scale, whereby '3' reflects the negative extreme on the Likert scale. The global score is generated by summing up all seven component scores and ranges from 0 to 21, with higher values corresponding to reduced sleep quality.
* Consequently, patients will be randomized to one of two groups: one group with general anesthesia maintenance based on an intravenous agent (propofol) and a second group with general anesthesia maintenance based on an inhalational agent (desflurane)
* Patients will be assessed postoperatively with sleep diaries regarding potential sleep disturbances while they will be subjected to a long-term assessment of sleep quality by the use of the PSQI one and three months postoperatively
* Since anesthetic-related differences in hormone profiles are expected, markers related to the neuroendocrine response to stress (cortisol, prolactin) will also be assessed to investigate differences between the two different anesthetic regimes
* Impaired melatonin secretion has been proposed as one of the mechanisms involved in postoperative sleep disturbances. It is therefore expected that different methods of anesthetic maintenance may affect the endogenous circadian melatonin rhythm in a different way. Consequently, melatonin secretion will also be measured to investigate potential desynchronization of melatonin rhythm as well as differences in melatonin secretion between the two different anesthetic techniques
* The clinical implications of this study lie in the fact that postoperative sleep disturbances can lead to postoperative hemodynamic instability, episodic hypoxemia and mental status deterioration, which can all untowardly affect the short and long-term postoperative outcome. It would be interesting to determine whether one of the two anesthetic regimes is superior to the other as far as postoperative disturbances in sleep architecture are concerned

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, American Society of Anesthesiologists (ASA) distribution I-III, scheduled for elective upper major abdominal surgery

Exclusion Criteria:

* Alcoholism
* Mental disability
* Psychiatric disease (depression, dementia)
* Preoperative use of sleeping medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
change from preoperative status of subjective sleep quality (evaluated by Pittburgh Sleep Quality Index) at one month postoperatively | preoperative status, one month postoperatively

SECONDARY OUTCOMES:
sleep diary | first postoperative week
cortisol levels | within the first 24 hours postoperatively
prolactin levels | within the first 24 hours postoperatively
melatonin levels | within the first 48 hours postoperatively
change from preoperative status of subjective sleep quality (evaluated by Pittburgh Sleep Quality Index) at three months postoperatively | preoperative status, three months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DEAA, Principal Investigator — Aretaieion University Hospital; Matthaios Stamelos, MD, Principal Investigator — Aretaieion University Hospital; Eriphylli Argyra, PhD, Study Chair — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Background] Rosenberg-Adamsen S, Kehlet H, Dodds C, Rosenberg J. Postoperative sleep disturbances: mechanisms and clinical implications. Br J Anaesth. 1996 Apr;76(4):552-9. doi: 10.1093/bja/76.4.552. No abstract available. PMID 8652329
- [Background] Knill RL, Moote CA, Skinner MI, Rose EA. Anesthesia with abdominal surgery leads to intense REM sleep during the first postoperative week. Anesthesiology. 1990 Jul;73(1):52-61. doi: 10.1097/00000542-199007000-00009. PMID 2360740
- [Background] Steinmetz J, Holm-Knudsen R, Eriksen K, Marxen D, Rasmussen LS. Quality differences in postoperative sleep between propofol-remifentanil and sevoflurane anesthesia in infants. Anesth Analg. 2007 Apr;104(4):779-83. doi: 10.1213/01.ane.0000255694.00651.5b. PMID 17377082
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Richardson J, Sabanathan S, Shah RD. Neuroendocrine response to mid and upper abdominal surgery. Acta Anaesthesiol Scand. 1997 Mar;41(3):433-4. doi: 10.1111/j.1399-6576.1997.tb04715.x. No abstract available. PMID 9113194
- [Background] Bourne RS, Mills GH. Melatonin: possible implications for the postoperative and critically ill patient. Intensive Care Med. 2006 Mar;32(3):371-9. doi: 10.1007/s00134-005-0061-x. Epub 2006 Feb 14. PMID 16477412
- [Background] Dispersyn G, Pain L, Touitou Y. Propofol anesthesia significantly alters plasma blood levels of melatonin in rats. Anesthesiology. 2010 Feb;112(2):333-7. doi: 10.1097/ALN.0b013e3181c920e2. PMID 20098135
- [Background] Lehmkuhl P, Prass D, Pichlmayr I. General anesthesia and postnarcotic sleep disorders. Neuropsychobiology. 1987;18(1):37-42. doi: 10.1159/000118390. PMID 3444524